CLINICAL TRIAL: NCT06376591
Title: Assessing the Efficacy of Different Carrier Systems in Oral Vitamin B12 Supplementation in Improving Circulatory B12 Levels in Healthy Adults
Brief Title: Assessing the Efficacy of Different Carrier Systems in Oral Vitamin B12 Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental Medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: No. LUMHS/REC/-291
Record Dates: First submitted 2024-04-12; First posted 2024-04-19 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-04

CONDITIONS: Vitamin B 12 Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Sucrosomial® B12 (Center 1) (Experimental): Participants will receive an oral single dose of 1000 mcg Sucrosomial® B12 supplement for 7 days.
  Interventions: Dietary Supplement: Vit B12
- B-SUB® B12 (Center 1) (Active Comparator): Participants will receive oral single dose of 1000 mcg B-SUB® B12 supplement for 7 days.
  Interventions: Dietary Supplement: Vit B12
- Sucrosomial® B12 (Center 2) (Experimental): Participants will receive an oral single dose of 1000 mcg Sucrosomial® B12 supplement for 7 days.
  Interventions: Dietary Supplement: Vit B12
- Mecogen SL® B12 (Center 2) (Active Comparator): Participants will receive an oral single dose of 1000 mcg Mecogen SL® B12 supplement for 7 days.
  Interventions: Dietary Supplement: Vit B12
- Sucrosomial® B12 (Center 3) (Experimental): Participants will receive an oral single dose of 1000 mcg Sucrosomial® B12 supplement for 7 days.
  Interventions: Dietary Supplement: Vit B12
- Evermin® B12 (Center 3) (Active Comparator): Participants will receive an oral single dose of 1000 mcg Evermin® B12 supplement for 7 days.
  Interventions: Dietary Supplement: Vit B12
- Neuromax® B12 (Center 3) (Active Comparator): Participants will receive an oral single dose of 1000 mcg Neuromax® B12 supplement for 7 days.
  Interventions: Dietary Supplement: Vit B12

INTERVENTIONS:
Dietary Supplement: Vit B12 — Sucrosomial® B12
  Arms: Sucrosomial® B12 (Center 1); Sucrosomial® B12 (Center 2); Sucrosomial® B12 (Center 3)
Dietary Supplement: Vit B12 — B-SUB® B12
  Arms: B-SUB® B12 (Center 1)
Dietary Supplement: Vit B12 — Mecogen SL® B12
  Arms: Mecogen SL® B12 (Center 2)
Dietary Supplement: Vit B12 — Evermin® B12
  Arms: Evermin® B12 (Center 3)
Dietary Supplement: Vit B12 — Neuromax® B12
  Arms: Neuromax® B12 (Center 3)

SUMMARY:
Vitamin B12, a vital nutrient, plays a crucial role in red blood cell formation, neurological function, and DNA synthesis. Deficiency in B12 can lead to anemia, neurological symptoms such as tingling or numbness, and cognitive impairment. Oral B12 supplementation serves as an effective strategy to address B12 deficiency, especially for individuals with limited dietary intake or absorption issues. Regular B12 supplementation can help restore body B12 levels, alleviate deficiency-related symptoms, and support overall health and well-being.

DETAILED DESCRIPTION:
The carrier system in oral vitamin B12 supplements plays a pivotal role in ensuring the stability and efficacy of the supplement. It helps protect the vitamin from degradation in the acidic environment of the stomach, enhancing its bioavailability. Additionally, the carrier system facilitates the transport of vitamin B12 across the gastrointestinal tract, promoting optimal absorption. By optimizing the delivery of B12 to the small intestine, the carrier system maximizes its potential for absorption into the bloodstream. Overall, the choice of carrier system significantly impacts the effectiveness of oral B12 supplementation in addressing deficiency and improving health outcomes.

Limited research exists regarding the exploration of various carrier systems used in oral B12 supplementation. This gap hinders a comprehensive understanding of how different carriers affect B12 absorption and efficacy. Further studies are needed to elucidate the optimal carrier system for maximizing B12 bioavailability and improving clinical outcomes. Expanding research in this area can enhance our knowledge and guide the development of more effective oral B12 supplements.

This study aims to compare the efficacy of sucrosomial and non-sucrosomial carrier systems in delivering vitamin B12 orally. By assessing absorption kinetics and clinical outcomes, we seek to determine the superiority of the sucrosomial carrier system in enhancing B12 bioavailability. Insights from this research could help in the development of more effective oral B12 supplements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, male or female, Aged 18 to 45 years
* Stable medical conditions, including stable cardiovascular, renal, hepatic, and hematological status,
* Normal vital signs Body mass index (BMI) 18-30 kg/m2
* Suboptimal vitamin B12 status, defined as serum B12 levels within the lower end of the reference range established by the laboratory conducting the assay.
* Willing and able to provide informed written consent.
* Able to comply with study procedures and follow-up visits as outlined in the protocol.

Exclusion Criteria:

* Known hypersensitivity or allergy to vitamin B12 or any of its components
* Known history of cobalt allergy or sensitivity.
* Severe malabsorption syndromes, including pernicious anemia or intestinal disorders affecting vitamin B12 absorption
* History of gastric bypass surgery or other procedures that significantly alter gastrointestinal anatomy or function
* Significant renal impairment (eGFR < 30 mL/min/1.73m²) or hepatic impairment
* Cancer
* Uncontrolled or significant cardiovascular disease, including recent myocardial infarction, unstable angina, or heart failure
* History of psychiatric illness or cognitive impairment that may impair their ability to comply with study procedures or provide informed consent
* Currently enrolled in another clinical trial involving investigational products or interventions.
* Pregnant or breast-feeding women
* Current use of acetaminophen, or nonsteroidal anti-inflammatory drugs, antibiotics, antacids, PPIs, multivitamins, or nutritional supplements with Vit B12
* Any other medical condition or circumstance that, in the investigator's judgment, would compromise the safety of the participant or the integrity of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Supplementation effect on circulatory vitamin B12 levels | Day 1, Day 3, Day 5, Day 7
  Changes in serum vitamin B12 levels

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Effects | one-week
  Number of participants report treatment-emergent adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat University of Medical and Health Sciences, Jamshoro, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Memon NM, Conti G, Brilli E, Tarantino G, Chaudhry MNA, Baloch A, Shafiq A, Mumtaz SU, Qaisar W, Iqtadar S, Abrar S, Kanwal A, Akhtar MH, Latif H, Rabbani F, Ujjan ID, Turroni S, Khan A. Comparative bioavailability study of supplemental oral Sucrosomial (R) vs. oral conventional vitamin B12 in enhancing circulatory B12 levels in healthy deficient adults: a multicentre, double-blind randomized clinical trial. Front Nutr. 2024 Nov 8;11:1493593. doi: 10.3389/fnut.2024.1493593. eCollection 2024. PMID 39582666